CLINICAL TRIAL: NCT00671892
Title: Role of TLR4 in Environmental Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Sundy (Other)
Responsible Party: Sponsor-Investigator, John Sundy, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3030-07-8R5; 12496-CP-007 (Other: NIEHS)
Record Dates: First submitted 2008-05-02; First posted 2008-05-05 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Asthma
Keywords: LPS endotoxin; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Challenge (Experimental): Experimental Challenge Challenge 1 saline 5000EU 10,000EU 20,000EU
  Challenge 2 Saline 40,000EU 80,000EU
  Interventions: Biological: Lipopolysaccharide endotoxin

INTERVENTIONS:
Biological: Lipopolysaccharide endotoxin — Delivered in nebulized form expressed in activity units(endotoxin units -EU).
  Subjects receive each dose 30 min after completing the previous dose, dose duration is approximately 10 minutes:
  Challenge One first saline then 5000 EU 10,000 EU 20,000 EU
  Challenge 1 and 2 must be at least 2 weeks apart.
  Challenge 2 Saline 40,000 EU 80,000 EU
  Other Names: (CCRE)LPS endotoxin from E. Coli 0:113 maintained by NIH

SUMMARY:
The overall goal of this project is to identify genes that are involved in the development of airflow obstruction and airway inflammation in asthmatics, and to determine whether polymorphisms in these differentially expressed genes predispose individuals to develop asthma. In this project, we hypothesize that polymorphisms of genes expressed by the airway epithelia in asthmatics following specific airway challenges predispose individuals to the development of asthma.

DETAILED DESCRIPTION:
The overall goal of this project is to identify genes that are involved in the development of airflow obstruction and airway inflammation in asthmatics, and to determine whether polymorphisms in these differentially expressed genes predispose individuals to develop asthma. Asthma is a complex genetic disorder that is caused by a number of unique gene-gene and gene-environment interactions. The search for asthma susceptibility genes has been complicated by the broad clinical phenotype of asthma, the polygenic inheritance pattern of this disease, and the substantial role of environmental exposures in the development and progression of asthma. Inhaled environmental agents induce several biologic responses in asthmatics; including the induction of acquired and innate immunity that leads to acute and chronic forms of airway inflammation and airway remodeling. Acquired immune responses to protein antigens, such as house dust mite allergen, often induce type 2 T lymphocyte-driven responses (Th2) which appear to be important in atopic asthma. Recent studies by our group and others demonstrate that innate immunity, initiated by inhalation of bacterial and viral pathogens, organic dusts, endotoxin or lipopolysaccharide (LPS), air pollution particulate matter, and ozone, can also cause acute and chronic forms of airflow obstruction, airway inflammation, and even airway remodeling. Emerging evidence indicates that both acquired and innate immune responses in the lung may be influenced by polymorphic genes. For instance, functional polymorphisms in the IL-4 receptor gene are thought to preferentially stimulate acquired Th2 immune responses to inhaled allergens, and we have recently shown that common co-segregating mutations in TLR4 (a transmembrane receptor for LPS) are associated with diminished airway responsiveness to inhaled LPS. These observations suggest that environmental challenges can be used to narrow the phenotype of asthma and investigate genetic susceptibility in biologically specific forms of asthma.

In this project, we hypothesize that polymorphisms of genes expressed by the airway epithelia in asthmatics following specific airway challenges predispose individuals to the development of asthma. To test this hypothesis, we plan to identify the genes that are differentially expressed by airway epithelial cells following challenge with stimuli that induce acquired (house dust mite) or innate (LPS) immune responses, and then determine whether polymorphisms in these genes are associated with the development of asthma in a separate, well characterized, familial cohort of asthmatics. This is a powerful approach that is designed to identify novel genes that are associated with both asthma pathogenesis (differentially expressed in the exposure-response study) and asthma susceptibility (genetically associated with asthma in a linkage/association study).

We hypothesize that individuals with the co-segregating Asp299Gly and Thr399Ile mutations in the TLR4 gene will exhibit a defective immune response to LPS, and that specific components of altered immunity in these individuals are linked to characteristic airway responses to LPS.

Specific Aim 1: Approximately 1000 individuals will be genotyped in order to establish 3 study groups: 10 subjects homozygous for the TLR4 299/399 mutation; 10 subjects heterozygous for the TLR4 299/399 mutation; and 10 subjects homozygous for wild type TLR 4.

Specific Aim 2: Ten individuals with wild type TLR4, 10 individuals heterozygous for mutant TLR4 and 10 individuals homozygous for mutant TLR4 will be phenotyped for airway responsiveness to inhaled LPS.

Specific Aim 3: In vitro immune responses to LPS will be measured in peripheral blood monocytes and PMNs from 10 individuals with wild type TLR4, 10 individuals heterozygous for mutant TLR4 and 10 individuals homozygous for mutant TLR4.

Specific Aim 4: The in vivo immune response to inhaled LPS will be assessed in bronchoalveolar lavage (BAL) fluid and cells, and airway endobronchial brush biopsy cells in 10 individuals with wild type TLR4, 10 individuals heterozygous for mutant TLR4 and 10 individuals homozygous for mutant TLR4.

ELIGIBILITY:
Inclusion Criteria:

* vital signs within normal limits
* negative methacholine challenge (non asthmatic)
* normal PFT's, CXR, EKG
* negative allergy skin tests (non atopic)
* never cigarette smoker
* no chronic illness
* no daily meds except contraceptives
* able and willing to sign informed consent
* not an employee working for,or a student under the authority of the PI's

Exclusion Criteria:

* allergic rhinitis past or present
* chronic illness resulting in altered lung function
* chronic daily medications
* cigarette smoking
* allergy to acetaminophen or albuterol
* pregnant or nursing females
* PFT results below cut off
* Positive allergy skin test
* Abnormal CXR or EKG
* Positive methacholine challenge
* Infection in the previous 2 weeks
* Past or present allergen immunotherapy
* Occupational exposure to hay or grain
* Other medical or psychological conditions which, in the opinion of the PI, may create undue risk to the subject or interfere with the subject's ability to comply with protocol requirements.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 855 (Actual)
Dates: Start 2001-09; Primary Completion 2006-08 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Ascertain individuals homozygous, and heterozygous for mutant TLR4 genotype, along with wild types by recruitment of healthy screening subjects in the community. | completed

SECONDARY OUTCOMES:
Assess the effect of TLR4 genotype on LPS endotoxin induced immune responses and assess the association of the LPS-induced immune response with LPS-induced airway responses. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: John S Sundy, M.D., PhD., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States